CLINICAL TRIAL: NCT05634018
Title: Prospective Assessment of the Biomechanical Properties of the Wall of an Aneurysmal-altered Abdominal Aorta According to the Results of in Vivo Ultrasound and an Associated Study of Strength Characteristics in Vitro
Brief Title: Comparison of the Biomechanical Properties of the Wall of an Aneurysmal-altered Abdominal Aorta According to the Results of in Vivo Ultrasound and an Associated Study of Strength Characteristics in Vitro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Other Study IDs: NRICP 22/11/22
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: the Strength Properties of the Aorta in Vivo; the Strength Properties of the Aorta in Vitro; Regression Model of Aortic Strength Properties in Vitro and in Vitro
Keywords: aneurysm wall strength; speckle tracking; shear yield strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: aneurysmectomy with sampling of a segment of the aneurysm wall — Patients with aneurysms of the abdominal aorta undergo an ultrasound examination of the abdominal aorta to assess the elastic properties of the aortic wall. The accessible wall of the abdominal aortic aneurysm is taken intraoperatively.
  In in vitro studies, the strength properties of the aneurysm wall are measured during uniaxial tension on a tensile testing machine, which makes it possible to evaluate the elastic properties of the test sample.
  The assessment of the boundaries of the linearity of the surface under study, as well as the yield strength of the vascular wall and thrombotic masses, is evaluated under shear stresses using a rheometer. To correlate the mechanical properties with the structural composition of the aneurysm tissue, spectral analysis of the studied tissues by laser-induced fluorescence and histological examination with staining of the obtained sections for the presence of elastic fibers, fibrous tissues and calcification will be used.

SUMMARY:
Identification of the regression model between the strength properties of tissue and its ultrasonic spectral characteristics.

DETAILED DESCRIPTION:
Patients with identified aneurysms of the abdominal aorta, who are planned for surgical treatment, undergo an ultrasound examination of the abdominal aorta to assess the elastic properties of the aortic wall using ultrasound speckle tracking. Intraoperatively, the accessible wall of the abdominal aortic aneurysm with a size of at least 10 cm2 is taken. and a section of the thrombotic cup of the aorta with a volume of up to 5 cm3. Pathologically altered tissues extracted for research are subject to removal during a standard operation for prosthetics of the infrarenal aorta and have no clinical significance for the patient.

In in vitro studies, the strength properties of the aneurysm wall are measured under uniaxial tension on a tensile testing machine, which makes it possible to evaluate the elastic properties of the test sample and obtain such parameters as Young's modulus (slope of the strain-stress diagram in a linear section at small deformations), as well as limiting strain values and loading.

The evaluation of the linearity boundaries of the surface under study, as well as the yield strength of the vascular wall and thrombotic masses, is evaluated under shear stresses using a rheometer. The tests will be carried out using special ground plane-to-plane instruments. To correlate the mechanical properties with the structural composition of the aneurysm tissue, spectral analysis of the tested tissues using the laser-induced fluorescence method and histological examination by staining the obtained sections for elastic fibers, fibrous tissues and calcification will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an aneurysmal expansion of the abdominal aorta who are indicated for surgery.
* Patients who consented to participate in this study

Exclusion Criteria:

* Chronic heart failure III-IV functional class according to the NYHA classification;
* Chronic decompensated "pulmonary" heart;
* Severe hepatic or renal insufficiency (bilirubin > 35 mmol / l, glomerular filtration rate < 60 ml / min);
* Polyvalent drug allergy;
* Malignant oncological diseases in the terminal stage with a predicted lifespan of up to 6 months;
* Acute violation of cerebral circulation;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged 45 to 75 with a diagnosed aneurysmal dilatation of the abdominal aorta requiring its surgical correction, recruited in accordance with the inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Calculate the relationship between the strength properties of the tissue and its ultrasonic spectral characteristics | 1 year
  Identification of the regression relationship between the elasto-elastic and strength properties of the tissue and its ultrasonic characteristics will make it possible to determine the most significant diagnostic ultrasonic criteria for aortic wall deformation, which determine the increased risk of its rupture and thromboembolic complications in a particular patient.

SECONDARY OUTCOMES:
Measurement of elastic-elastic properties of the aortic wall using ultrasonic speckle tracking | at least one day prior to surgery
  Patients with identified aneurysms of the abdominal aorta, who are planned for surgical treatment, undergo an ultrasound examination of the abdominal aorta to assess the elastic properties of the aortic wall using ultrasound speckle tracking. with the construction of a graph of elastic deformation segment by segment
Measurement of the strength properties of the aneurysm wall in uniaxial tension in vitro | 1 month
  evaluate the elastic properties of the tested sample and obtain parameters such as Young's modulus (the slope of the strain-stress diagram in the linear section at small strains)
Measure linearity limits as well as shear yield strength in vitro | 1 month
  The evaluation of the linearity boundaries of the surface under study, as well as the yield strength of the vascular wall and thrombotic masses, is evaluated under shear stresses using a rheometer

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Alexander A Gostev, Novosibirsk, Novosibirskaya Obl
  - Federal State Institution Academician E.N.Meshalkin Novosibirsk State Research Institute Of Circulation Pathology Rusmedtechnology, Novosibirsk
  - E. Meshalkin National Medical Research Center, Novosibirsk

IPD SHARING:
Plan to Share IPD: Yes
Access to data after first publication at the request of researchers
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Access to data after first publication at the request of researchers
Access Criteria: on personal request